CLINICAL TRIAL: NCT02210897
Title: Influence of Renal Function on the Circadian Variation of Cardiac Troponin
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 14-2-016
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cardiac troponin is the preferred biomarker for the diagnosis of acute myocardial infarction. Whereas the diagnosis is based on an increase and/or decrease in the concentrations of cardiac troponins with at least one value above the 99th percentile value of the reference population together with the evidence of ischemia, serial sampling is needed. Knowledge of the variation in cardiac troponin levels over time in individuals in a normal rest state (not during an acute myocardial infarction), also called the biological variation, is important regarding the interpretation of the serial cardiac troponin levels. A recent study by our group showed a circadian rhythm in cardiac troponin levels. This circadian rhythm is important regarding the interpretation of the serial cardiac troponin levels.

Increased cTnI and cTnT concentrations are common in subjects with renal impairment. The mechanism of the elevated concentration of cTn in these subjects is still unclear. It is hypothesized that impaired renal clearance contributes to elevated levels of cTn. However, it is not clear whether renal function affects the biological variation and circadian rhythm of cTn. The monitoring of the biological variation and circadian rhythm of cTn in subjects with impaired renal function creates the opportunity to assess the effect of renal clearance on the circadian rhythm of cardiac troponins.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3 or 4
* No dialysis
* No evidence of active, acute cardiovascular disease

Exclusion Criteria:

* History of acute myocardial infarction in the last year
* History of pulmonary embolism in the last six months
* Anemia (Hb < 6.5 mmol/L)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic kidney disease (CKD) stage 3 and 4
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Cardiac Troponins (cardiac troponin I (cTnI) and cardiac troponin T (cTnT)) | up to three months

OTHER OUTCOMES:
24-hour automatic blood pressure measurements (diastolic and systolic blood pressure) | total time 25 hours (first testday)
Urine concentrations of creatinine, electrolytes and cardiac markers | every 4 hours, total time 25 hours (first testday)

CONTACTS AND LOCATIONS:
Overall Officials: Steven JR Meex, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Background] Klinkenberg LJ, van Dijk JW, Tan FE, van Loon LJ, van Dieijen-Visser MP, Meex SJ. Circulating cardiac troponin T exhibits a diurnal rhythm. J Am Coll Cardiol. 2014 May 6;63(17):1788-95. doi: 10.1016/j.jacc.2014.01.040. Epub 2014 Feb 26. PMID 24583293
- [Derived] Breidthardt T, van Doorn WPTM, van der Linden N, Diebold M, Wussler D, Danier I, Zimmermann T, Shrestha S, Kozhuharov N, Belkin M, Porta C, Strebel I, Michou E, Gualandro DM, Nowak A, Meex SJR, Mueller C. Diurnal Variations in Natriuretic Peptide Levels: Clinical Implications for the Diagnosis of Acute Heart Failure. Circ Heart Fail. 2022 Jun;15(6):e009165. doi: 10.1161/CIRCHEARTFAILURE.121.009165. Epub 2022 Jun 7. PMID 35670217